CLINICAL TRIAL: NCT06822699
Title: The Influence of Thirty-degree Leg Elevation on Noradrenaline Requirements Administered as a Prophylactic Variable Infusion During Cesarean Delivery: An Open Label Randomized Controlled Trial
Brief Title: The Influence of Leg Elevation on Noradrenaline Requirements During Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Adolf Helmy, lecture of anesthesia and critical care Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: leg elevation and noradrenalin
Record Dates: First submitted 2025-02-07; First posted 2025-02-12 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-03

CONDITIONS: Spinal Hypotension; Hypoperfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Leg elevation group (Experimental): leg will be elevated 30 degrees immediately after spinal anesthesia
  Interventions: Device: Leg elevation
- Control group (No Intervention): Legs will remain supine after spinal anesthesia

INTERVENTIONS:
Device: Leg elevation — leg will be raised 30 degrees after spinal anesthesia using standardized pillow
  Arms: Leg elevation group

SUMMARY:
Spinal anesthesia is a widely chosen technique in obstetric theaters due to several advantages, however sympathetic block results in hypotension that carry several consequences on maternal and fetal health, thus early prediction and management takes high priority. in this regards recent recommendations suggest the use of prophylactic vasopressors like noradrenaline, researchers of this study aimed to explore the impact of leg elevation on prophylactic noradrenaline dose

DETAILED DESCRIPTION:
after spinal anesthesia, patients will be randomly allocated into 2 groups : Leg elevation group and control group.

noradrenaline will be used as variable infusion starting from 0.05 microgram/kg/min up to 0.14 microgram /kg/minute.

noradrenaline infusion will be continued till delivery of the baby

ELIGIBILITY:
Inclusion Criteria:

* full term
* singleton pregnancy
* ASA II

Exclusion Criteria:

* decline to participate
* baseline SBP <100 mmHg
* failed spinal anesthesia
* allergy to local anesthetic
* coagulopathy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women undergoing elective ceserean section
Enrollment: 80 (Actual)
Dates: Start 2025-03-14 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Average noradrenaline requirements | baseline to delivery of the baby
  average noradrenaline requirements in both groups (mcg/kg/min)

SECONDARY OUTCOMES:
Total noradrenaline requirements | baseline to delivery
incidence of spinal hypotension | baseline to delivery
incidence of severe hypotension | baseline to delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available from corresponding author upon reasonable request

REFERENCES:
- [Background] Hasanin A, Aiyad A, Elsakka A, Kamel A, Fouad R, Osman M, Mokhtar A, Refaat S, Hassabelnaby Y. Leg elevation decreases the incidence of post-spinal hypotension in cesarean section: a randomized controlled trial. BMC Anesthesiol. 2017 Apr 24;17(1):60. doi: 10.1186/s12871-017-0349-8. PMID 28438121
- [Background] Lyu W, Zhang Z, Li C, Wei P, Feng H, Zhou H, Zheng Q, Zhou J, Li J. Intravenous initial bolus during prophylactic norepinephrine infusion to prevent spinal hypotension for cesarean delivery: A randomized controlled, dose-finding trial. J Clin Anesth. 2024 Oct;97:111562. doi: 10.1016/j.jclinane.2024.111562. Epub 2024 Jul 23. PMID 39047530
- [Background] Hasanin AM, Amin SM, Agiza NA, Elsayed MK, Refaat S, Hussein HA, Rouk TI, Alrahmany M, Elsayad ME, Elshafaei KA, Refaie A. Norepinephrine Infusion for Preventing Postspinal Anesthesia Hypotension during Cesarean Delivery: A Randomized Dose-finding Trial. Anesthesiology. 2019 Jan;130(1):55-62. doi: 10.1097/ALN.0000000000002483. PMID 30335625
- [Background] Kinsella SM, Carvalho B, Dyer RA, Fernando R, McDonnell N, Mercier FJ, Palanisamy A, Sia ATH, Van de Velde M, Vercueil A; Consensus Statement Collaborators. International consensus statement on the management of hypotension with vasopressors during caesarean section under spinal anaesthesia. Anaesthesia. 2018 Jan;73(1):71-92. doi: 10.1111/anae.14080. Epub 2017 Nov 1. No abstract available. PMID 29090733
- [Background] Yu C, Gu J, Liao Z, Feng S. Prediction of spinal anesthesia-induced hypotension during elective cesarean section: a systematic review of prospective observational studies. Int J Obstet Anesth. 2021 Aug;47:103175. doi: 10.1016/j.ijoa.2021.103175. Epub 2021 May 1. PMID 34034957
- [Derived] Helmy MA, Naguib NN, Helmy KA, Milad LM. The influence of thirty-degree leg elevation on noradrenaline requirements administered as a prophylactic variable infusion during cesarean delivery, an open-label randomized controlled trial. J Anesth Analg Crit Care. 2025 Oct 28;5(1):73. doi: 10.1186/s44158-025-00290-7. PMID 41152963